CLINICAL TRIAL: NCT01067313
Title: Evaluation of Continuous Hemodialysis With an Enhanced Middle Molecule Clearance Membrane in Intensive Care
Brief Title: Continuous Hemodialysis With an Enhanced Middle Molecule Clearance Membrane
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fresenius Medical Care France (Industry)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Professor Bernard Allaouchiche, Edouard Herriot Hospital, Lyon, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD-RE-01-F
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2010-02

CONDITIONS: Septic Shock
Keywords: Intensive Care Unit; continuous hemodialysis; continuous hemofiltration; High Cut-off membrane; "Enhanced middle molecule clearance" membrane; Septic shock; Acute kidney injury; Blood purification; Renal replacement therapy
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialyzer Ultraflux EMiC2 (Experimental): Dialyzer Ultraflux EMiC2 used in Continuous Hemodialysis
  Interventions: Device: Dialyzer Ultraflux EMiC2
- Dialyzer Ultraflux AV1000S (Active Comparator): Dialyzer Ultraflux AV1000S used in continuous Hemofiltration
  Interventions: Device: Dialyzer Ultraflux AV1000S

INTERVENTIONS:
Device: Dialyzer Ultraflux EMiC2 — Dialysate flow rate = 40 ml/kg/h The treatment duration may be variable depending on modifications in patient health status, but will not exceed 3 sessions of 48 hours each.
  Arms: Dialyzer Ultraflux EMiC2
Device: Dialyzer Ultraflux AV1000S — Ultrafiltration flow rate = 40 ml/kg/h The blood flow rate will be adjusted to obtain a filtration fraction of 20%. Reinjection = 100% postdilution. The treatment duration may be variable depending on modifications in patient health status, but will not exceed 3 sessions of 48 hours each.
  Arms: Dialyzer Ultraflux AV1000S

SUMMARY:
This study aims to demonstrate equivalence in terms of molecule removal between continuous hemodialysis using an "enhanced middle molecule clearance" membrane(Ultraflux EMiC2) and continuous hemofiltration using a standard membrane (Ultraflux AV1000S) in ICU patients requiring continuous renal replacement therapy.

DETAILED DESCRIPTION:
In sepsis, the removal of middle molecular weight molecules such as cytokines (also called blood purification), has shown a great interest in intensive care during the last decades. Indeed, these cytokines are involved in the development of the multi-organ failure syndrome when patients are in septic shock. There is some evidence to suggest that extracorporeal therapies (hemofiltration-hemodialysis)are interesting tools to modulate the inflammatory response and to restore the immune homeostasis.

However, hemodialysis using "conventional" membranes does not allow the removal of middle molecules. Conversely, high-volume hemofiltration is an appropriate therapy but it has a lot of drawbacks due to the high ultrafiltration rates (removal of beneficial small molecules, technical and economical issues due to the use of large amounts of fluid replacement). Finally, high cut-off hemofiltration has been reported to be associated with significant albumin loss.

Therefore, continuous "enhanced middle molecule clearance" hemodialysis could be an interesting alternative, making possible the removal of these middle molecules without significant albumin loss and with some theoretical advantages (reduced cost due to the possibility to produce the dialysate from a water circuit, decreased nursing workload).

The aim of this study is to assess the clearances of different kind of molecules (small, middle and large) when continuous enhanced middle molecule clearance hemodialysis is applied to septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years.
* ICU patients with septic shock and AKI requiring continuous renal replacement.
* Patient able to agree to be enrolled in the study with informed consent. If the patient can not provide consent, only the consent of family members will be sought if they are present and, to default, the opinion of trustworthy person under article L.1111-6 of the French Health Code. If there is no family present, or trustworthy person designated, the subject will not be included in the study.

Exclusion Criteria:

* Pregnancy or lactation.
* Participation in another research protocol.
* People particularly vulnerable as defined in Articles L.1121-5, L.1121-6, L.1121-7, L.1121-8 et L.1122-1-2 of the French Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Clearance of Urea | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Clearance of creatinine | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Clearance of total protein | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Clearance of albumin | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Clearance of Beta 2-microglobulin | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Free light chains kappa of Immunoglobulins | At 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours

SECONDARY OUTCOMES:
Mean arterial pressure | Before connecting Patient and at 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
vasopressor requirement | Before connecting Patient and at 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
PaO2 / FiO2 | Before connecting Patient and at 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Heart rate | Before connecting Patient and at 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours
Lactate level | Before connecting Patient and at 15 minutes, 60 minutes, 4 hours, 12 hours, 24 hours and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Allaouchiche, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Edouard Herriot Hospital, P Reanimation, Lyon, France